CLINICAL TRIAL: NCT04768660
Title: The Use of Non-pharmacological Agent to Accelerate Gastrointestinal Recovery in Patients Undergoing Pancreatic Head Resection
Brief Title: Effects of Chewing Gum Against Postoperative Ileus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Mokbel, andrew mokbel mahani sawers, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: chewing gum postoperative
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-09

CONDITIONS: Pancreas Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Chewing Gum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- normal (Other): people will not use chewing gums after whipple operation
  Interventions: Other: gum

INTERVENTIONS:
Other: gum — Other: Chewing gum ChiczaTM organic chewing gum 6 pieces a day Other: Glucose 12ml glucose solution (13,6g) per day

SUMMARY:
The purpose of this study is to determine whether the use of chewing gum effects postoperative ileus after pancreaticoduodenectomy

DETAILED DESCRIPTION:
Postoperative ileus is common after surgery. One non-pharmacological intervention that has shown promising results in reducing the duration of postoperative ileus is chewing gum after surgery. However, this has not been investigated in upper gastrointestinal surgery such as pancreatic surgery. Hence the aim of this study was to investigate the effects of chewing gum treatment on patients undergoing pancreaticoduodenectomy due to pancreatic or periampullary cancer.

This study was conducted as a phase-III trial. Patients diagnosed with pancreatic tumours scheduled for pancreaticoduodenectomy were included. The treatment group received chewing gum postoperatively and standard care. Controls received glucose solution and standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Pancreatic or periampullary cancer and scheduled to undergo pancreaticoduodenectomy.

Exclusion Criteria:

* 2. Ongoing treatment for mental disease 3. Diagnosed neurological injuries or diseases affecting the ability to swallow or gastric function 4. Ongoing abuse of alcohol or other drugs 5. Previously known allergies to the content of chewing gum 6. Additional surgery after primary surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02-14 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
First flatus after surgery | (with in the first 21 days)
  From day of surgery until first postoperative flatus
Length of hospital stay | (with in the first 21 days) ]
  Time Frame: From day of surgery until discharge from surgical ward

IPD SHARING:
Plan to Share IPD: Undecided